CLINICAL TRIAL: NCT00811928
Title: A Randomized, Open Label Parallel Controlled, Multicenter Study to Evaluate Safety and Efficacy of Posaconazole Oral Suspension Vs. Fluconazole (Capsule) in High-risk Leukopenic Patients for Prevention of Invasive Fungal Infection
Brief Title: Safety and Efficacy Study of Posaconazole vs. Fluconazole for Prevention of Invasive Fungal Infection (P05387 AM1)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P05387
Record Dates: First submitted 2008-12-18; First posted 2008-12-19 (Estimated); Results first posted 2011-09-13 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-03

CONDITIONS: Leukopenia
Keywords: high-risk leukopenic patients
MeSH Terms: conditions — Leukopenia | interventions — posaconazole; Fluconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Posaconazole (Active Comparator): Posaconazole oral suspension 200 mg three times a day (TID)
  Interventions: Drug: Posaconazole
- Fluconazole (Active Comparator): Fluconazole 400 mg once daily (QD)
  Interventions: Drug: Fluconazole

INTERVENTIONS:
Drug: Posaconazole — 40 mg/mL; 200 mg (5 mL) TID
  Treatment was continued with each cycle of chemotherapy until:
  * The onset of a proven or probable diagnosis of invasive fungal infection (IFI)
  * 3 chemotherapy cycles or
  * Total treatment duration up to 12 weeks (84 days)
  Other Names: Noxafil; SCH 056592
  Arms: Posaconazole
Drug: Fluconazole — 50 mg/capsule (2 capsules), 150 mg/capsule (2 capsules);
  400 mg QD
  Treatment was continued with each cycle of chemotherapy until:
  * The onset of a proven or probable diagnosis of invasive fungal infection (IFI)
  * 3 chemotherapy cycles or
  * Total treatment duration up to 12 weeks (84 days)
  Arms: Fluconazole

SUMMARY:
A randomized, open label parallel controlled, multicenter study to evaluate safety and efficacy of Posaconazole oral suspension vs Fluconazole (capsule) in high-risk leukopenic patients for prevention of invasive fungal infection

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 18-70 years of age of either sex
* Persistent neutropenia (Absolute Neutrophil Count [ANC] < 500/mm^3 [0.5x10^9/L]）or probable neutropenia in 3-5 days is anticipated. Neutropenia >= 7 days caused by the following reasons

  * Standard or dose-intense chemotherapy, anthracyclines or other acceptable chemotherapies ( any investigational drug is not permitted) for Acute Myelogenous Leukemia (AML) treatment
  * Retreatment of chemotherapy in case of AML recurrence
  * Myelodysplastic syndrome (MDS) shifts to AML and bone marrow arrest induction chemotherapy is required (not including acute phase of chronic myelogenous leukemia [CML])
* Informed consent obtained from participant or legal guardian

Exclusion Criteria:

* Participants previously treated with amphotericin B (AMB), fluconazole (FLZ), or itraconazole (ITZ) within 30 days of enrollment.
* Participants who have taken the following drugs:

  * terfenadine, cisapride, and ebastine within 24 hours before entry
  * astemizole at entry or within 10 days before entry
  * cimetidine, rifampin, carbamazepine, phenytoin, rifabutin, barbiturates, isoniazid atharanthine and anthracyclines within 24 hours before entry
* The above drugs are refrained during the investigation
* Serious organ diseases except hematological disorder such as cardiac or neurologic disorders or impairment expected to be unstable or progressive during the course of this study (eg, seizures or demyelinating syndromes, acute myocardial infarction within 3 months of study entry, myocardial ischemia, congestive heart failure, atrial fibrillation with ventricular rate <60/min, or history of torsades de pointes, symptomatic ventricular or sustained arrhythmias), unstable electrolyte abnormalities.
* Participants who have used any investigational drugs or biologic agents other than their chemotherapy regimens within 30 days of study entry.
* Prior enrollment in this study.
* Participants with known or suspected hypersensitivity or idiosyncratic reaction to azole agents or amphotericin B.
* Participants with known or suspected invasive fungal infection (IFI) at screen
* Participants with severe renal insufficiency (estimated creatinine clearance less than 50 mL/minute or likely to require dialysis during the study), Alanine transaminase (ALT), Aspartate transaminase (AST), alkaline phosphatase or total bilirubin are >2× (Upper Limit of Normal) ULN.
* Participants having an electrocardiogram (ECG) with a prolonged QTc interval: QTc greater than 450 msec for men and greater than 470 msec for women.
* Participants with AML or CML history.
* Participants with a history of allogeneic hematopoietic stem cell, bone marrow transplantation, autologous stem cell transplantation history.
* Female participants who are pregnant or are nursing.
* Alcohol and/or drug abuse.
* Participants cannot be compliant in the opinion of the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2008-11; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Shen Y, Huang XJ, Wang JX, Jin J, Hu JD, Yu K, Wu DP, Wang SJ, Yu L, Chen XQ, Liu T, Liang YM, Chen FP, Li Y, Shen ZX. Posaconazole vs. fluconazole as invasive fungal infection prophylaxis in China: a multicenter, randomized, open-label study. Int J Clin Pharmacol Ther. 2013 Sep;51(9):738-45. doi: 10.5414/CP201880. PMID 23924680

RESULTS

PARTICIPANT FLOW:
Groups:
- Posaconazole: Posaconazole oral suspension (40 mg/ml), 200 mg (5mL) three times a day (TID) with meals
- Fluconazole: Fluconazole 400 mg daily (QD), given as 2 capsules of 50 mg and 2 capsules of 150 mg (a total of 4 capsules) with or without food
Period: Overall Study
Arm/Group | Posaconazole | Fluconazole
Started | 129 | 123
Completed | 90 | 90
Not Completed | 39 | 33
Not completed — AEs and SAEs Including Death | 7 | 11
Not completed — Withdrawal by Subject | 18 | 12
Not completed — Did Not Take Study Drug | 3 | 0
Not completed — Without Primary Efficacy Endpoint Data | 7 | 4
Not completed — Investigator Decision | 2 | 1
Not completed — Poor Compliance | 2 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Posaconazole | Fluconazole | Total
Number analyzed (Participants) | 117 | 117 | 234
Age, Continuous [Mean (Standard Deviation); unit: participants] — The full analysis set (FAS) included all of those randomized participants who received at least one dose of study drug, and had at least one post-treatment follow-up data of primary efficacy variable.
  participants | 39.3 (13.01) | 40.6 (12.50) | 40.4 (12.73)
Sex: Female, Male [Count of Participants; unit: Participants] — The full analysis set (FAS) included all of those randomized participants who received at least one dose of study drug, and had at least one post-treatment follow-up data of primary efficacy variable.
  Participants
    Female | 62 | 65 | 127
    Male | 55 | 52 | 107

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Proven or Probable Diagnosis of Invasive Fungal Infection (IFI) During the Treatment Period
Description: Number of participants developing a proven or probable IFI from randomization to the last dosage date (up to 12 weeks [84 days]) plus 7 days. IFI diagnosis criteria may include: persistent fever, failure of appropriate broad-spectrum antibiotic treatment concomitant with lower respiratory tract infection symptoms, microbiological criteria with corresponding clinical signs and symptoms.
Time Frame: Up to 12 Weeks (84 days) plus 7 days
Population: The full analysis set (FAS) included all of those randomized participants who received at least one dose of study drug, and had at least one post-treatment follow-up data of primary efficacy variable.
Measure: Number; unit: participants
Arm/Group | Posaconazole | Fluconazole
Number analyzed (Participants) | 117 | 117
participants | 4 | 11
Statistical Analysis 1: Comparison: Posaconazole vs Fluconazole; Test type: Non-Inferiority or Equivalence — The upper limit of the 95% Confidence Interval for the difference in incidence defined as (# of participants affected with proven or probable IFI/ # of participants in the FAS population at risk)*100% (posaconazole minus fluconazole) had to be < 4 in order to be considered non-inferior. IFI occurred: proven+probable; Difference for the incidence = -5.88, 95% CI 2-sided [-12.21 to 0.25] — Posaconazole minus fluconazole

2. Secondary Outcome: Number of Participants With Proven or Probable Diagnosis of IFI Within 100 Days From Randomization
Description: Number of participants who developed a proven or probable IFI from randomization date to Day 100 of follow-up visit. IFI diagnosis criteria may include: persistent fever, failure of appropriate broad-spectrum antibiotic treatment concomitant with lower respiratory tract infection symptoms, microbiological criteria with corresponding clinical signs and symptoms.
Time Frame: From randomization date to Day 100
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Posaconazole | Fluconazole
Number analyzed (Participants) | 117 | 117
participants | 5 | 16
Statistical Analysis 1: Comparison: Posaconazole; Test type: Superiority or Other; Percentage of Participants = 4.27, 95% CI 2-sided [1.4 to 9.7] — IFI Incidence for the Posaconazole group = (# of participants affected with proven or probable IFI/ # of participants in the FAS population at risk)*100%
Statistical Analysis 2: Comparison: Fluconazole; Test type: Superiority or Other; Percentage of Participants = 13.68, 95% CI 2-sided [8.0 to 21.3] — IFI Incidence for the Fluconazole group = (# of participants affected with proven or probable IFI/ # of participants in the FAS population at risk)*100%

3. Secondary Outcome: Time From Randomization to the First Onset of Proven or Probable IFI
Description: The time measured in days to the first occurrence of proven/probable IFI diagnosis in the entire FAS population from randomization to Day 100 of follow-up visit. Participants may not have accepted immediate antifungal treatment and later received antifungal treatment based upon further investigator review of the participant's IFI condition. IFI diagnosis criteria may include: persistent fever, failure of appropriate broad-spectrum antibiotic treatment concomitant with lower respiratory tract infection symptoms, positive blood/biopsy cultures with corresponding clinical signs and symptoms.
Time Frame: From randomization date to Day 100
Population: as for outcome 1
Measure: Number; unit: Days
Arm/Group | Posaconazole | Fluconazole
Number analyzed (Participants) | 117 | 117
Days | 8 | 2

4. Secondary Outcome: Time From Randomization to Administration of First Systemic Antifungal Intravenous (IV) Therapy
Description: The time measured in days from randomization to the administration of the first concomitant systemic anti-fungal therapy in the entire FAS population. Not all participants who accepted systemic anti-fungal therapy may have had a IFI clinical diagnosis. IFI diagnosis criteria for antifungal therapy administration may include: persistent fever, failure of appropriate broad-spectrum antibiotic treatment concomitant with lower respiratory tract infection symptoms, microbiological criteria with corresponding clinical signs and symptoms.
Time Frame: Up to 12 weeks (84 days)
Population: as for outcome 1
Measure: Number; unit: Days
Arm/Group | Posaconazole | Fluconazole
Number analyzed (Participants) | 117 | 117
Days | 4 | 1

5. Secondary Outcome: Number of Participants With Clinical Failure During Treatment
Description: Clinical failure was defined as follows:
  * Presence of a proven or probable IFI
  * Systemic antifungal treatment (IV) for 4 consecutive days or more than 10 days total
  * Discontinuation due to adverse event (AE) possibly or probably related to study drug
  * Lost-to-follow-up or discontinuation from the study for any reason with loss to follow-up during the Treatment Phase
Time Frame: Up to 12 weeks (84 days)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Posaconazole | Fluconazole
Number analyzed (Participants) | 117 | 117
participants | 37 | 51
Statistical Analysis 1: Comparison: Posaconazole; Test type: Superiority or Other; Percentage of Participants = 31.62, 95% CI 2-sided [23.3 to 40.9] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Fluconazole; Test type: Superiority or Other; Percentage of Participants = 41.88, 95% CI 2-sided [32.8 to 51.4] — [estimate comment as in outcome 2, analysis 2]

6. Secondary Outcome: Number of Participants in Whom All-cause Mortality Occurred Within 100 Days From Randomization
Description: Death from any cause.
Time Frame: Randomization date to Day 100
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Posaconazole | Fluconazole
Number analyzed (Participants) | 117 | 117
participants | 3 | 8
Statistical Analysis 1: Comparison: Posaconazole; Test type: Superiority or Other; Percentage of Participants = 2.56, 95% CI 2-sided [0.5 to 7.3] — All-Cause Mortality Rate is the percentage of participants with mortality from any cause
Statistical Analysis 2: Comparison: Fluconazole; Test type: Superiority or Other; Percentage of Participants = 5.98, 95% CI 2-sided [2.4 to 11.9] — All-Cause Mortality Rate is the percentage of participants with mortality from any cause

7. Secondary Outcome: Number of Participants in Whom Mortality is Unlikely, Possibly, and Probably Related to Fungal Infection Occurred Within 100 Days From Randomization
Description: Exact Causes of Death and Their Relationship to IFI Episode Were As Follows:
  * Unlikely related: participant completed treatment and cause of death was due to primary disease or complication
  * Possibly related: IFI undergoing treatment without stabilization, or with failure to have a complete remission, where cause of death might have been due to IFI, including progression or relapse of primary disease
  * Probably related: autopsy or clinical signs suggested that progression of IFI was the probable cause of death
Time Frame: From randomization date to Day 100
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Posaconazole | Fluconazole
Number analyzed (Participants) | 117 | 117
participants | 0 | 0

ADVERSE EVENTS:
Time Frame: From screening to the last dosage date plus 30 days
Description: Safety analysis set (SS) included randomized participants who received at least one dose of study drug and had valid data of safety endpoints available for at least one follow-up visit after treatment.
Arm/Group | Posaconazole | Fluconazole
Serious Adverse Events (participants affected / at risk) | 7/124 | 10/121
Other Adverse Events (participants affected / at risk) | 82/124 | 81/121
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Posaconazole (N=124) | Fluconazole (N=121)
Bone marrow depression (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Death (General disorders) | 1 (1) | 2 (2)
Oedema (General disorders) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Cerebellar haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) — One participant developed an SAE of life-threatening Respiratory Failure due to Cerebral Infarction, in the AE tables it was counted as a Cerebral Infarction
Consciousness disturbance (Nervous system disorders) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cerebral haemorrhage (Vascular disorders) | 2 (2) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Posaconazole (N=124) | Fluconazole (N=121)
Bone marrow depression (Blood and lymphatic system disorders) | 7 (9) | 4 (6)
Abdominal discomfort (Gastrointestinal disorders) | 10 (15) | 5 (5)
Anal disorder (Gastrointestinal disorders) | 11 (12) | 14 (17)
Constipation (Gastrointestinal disorders) | 7 (8) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 15 (15) | 17 (18)
Gingivitis (Gastrointestinal disorders) | 19 (27) | 18 (19)
Mucosal inflammation (Gastrointestinal disorders) | 13 (13) | 12 (15)
Nausea (Gastrointestinal disorders) | 16 (20) | 15 (16)
Vomiting (Gastrointestinal disorders) | 7 (8) | 7 (7)
Chest discomfort (General disorders) | 4 (6) | 7 (7)
Pain (General disorders) | 7 (9) | 6 (6)
Pyrexia (General disorders) | 39 (61) | 39 (63)
Hepatic function abnormal (Investigations) | 25 (27) | 21 (29)
Electrolyte imbalance (Metabolism and nutrition disorders) | 20 (43) | 15 (29)
Dizziness (Nervous system disorders) | 7 (10) | 2 (2)
Headache (Nervous system disorders) | 9 (10) | 6 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 12 (22) | 6 (7)
ENT disorder (Respiratory, thoracic and mediastinal disorders) | 23 (31) | 20 (26)
Respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 17 (21) | 16 (20)
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 7 (8) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 19 (21) | 19 (23)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Principal Investigator agrees not to publish or publicly present any interim results of the Protocol study without the prior written consent of the SPONSOR. The Principal Investigator further agrees to provide to the

SPONSOR thirty (30) days prior to submission for publication or presentation, review copies of abstracts or manuscripts for publication that report any results of the Protocol study.